CLINICAL TRIAL: NCT05224180
Title: Obstructive Sleep Apnea in Never Smokers With Newly Diagnosed Lung Cancer: Prevalence and Impact on Prognosis
Brief Title: OSA in Never Smokers With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Assistant Professor, Seoul National University Hospital
Other Study IDs: 21071691236
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; Obstructive Sleep Apnea
MeSH Terms: conditions — Lung Neoplasms; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have yielded inconsistent findings regarding the association between obstructive sleep apnea and the prevalence and mortality of lung cancer. Smoking history, a common risk factor for lung cancer, chronic obstructive pulmonary disease, and obstructive sleep apnea, may act as a confounding variable, limiting interpretation of the results. The aim of this study is to evaluate the prevalence of obstructive sleep apnea in never smokers with lung cancer and to determine the effect of obstructive sleep apnea on the prognosis of lung cancer. Enrolled patients will undergo respiratory polygraphy before beginning treatment for lung cancer. This prospective cohort includes both cross sectional and longitudinal analyses.

ELIGIBILITY:
Inclusion Criteria:

- Never smokers who are admitted to the Seoul National University Hospital and newly diagnosed with lung cancer, with ECOG Performance Status 0 or 1

Exclusion Criteria:

* Patients who have received treatment for lung cancer before the enrollment
* Patients who have received treatment for OSA before the enrollment
* Patients with an expected life expectancy of less than 3 months
* Patients with neuromuscular disease, chronic opioid medication use, or severe insomnia not controlled by medication
* Patients receiving supplemental oxygen therapy due to underlying diseases including heart failure, chronic obstructive pulmonary disease, interstitial pulmonary disease, hypoventilation syndrome, stroke, or whose baseline oxygen saturation is less than 90%
* Patients with unstable medical conditions within the preceding 3 months (hospitalization due to acute exacerbation of underlying lung disease, diagnosis of unstable angina or myocardial infarction, history of percutaneous coronary intervention or coronary artery bypass surgery, or diagnosis of transient ischemic attack or stroke)
* Patients with an inability or unwillingness to provide informed consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients in a tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea in never smokers with lung cancer | 1 week
  A primary outcome measure in a cross-sectional analysis of a prospective cohort study
Effects of obstructive sleep apnea on lung cancer mortality and overall mortality | Follow up for 5 years
  A primary outcome measure in a longitudinal analysis of prospective cohort study

SECONDARY OUTCOMES:
Association between apnea-hyponea index (AHI) and the stage of lung cancer | 1 week
  A secondary outcome measure in a cross-sectional analysis of a prospective cohort study.
Association between the oxygen desaturation index (ODI) and the stage of lung cancer | 1 week
  A secondary outcome measure in a cross-sectional analysis of a prospective cohort study.
Association between the sleep time spent with oxygen saturation< 90% (TS90) and the stage of lung cancer | 1 week
  A secondary outcome measure in a cross-sectional analysis of a prospective cohort study.
Effect of the apnea-hyponea index (AHI) on lung cancer mortality and overall mortality | Follow up for 5 years
  A secondary outcome measure in a longitudinal analysis of prospective cohort study.
Effect of the oxygen desaturation index (ODI) on lung cancer mortality and overall mortality | Follow up for 5 years
  A secondary outcome measure in a longitudinal analysis of prospective cohort study.
Effect of the sleep time spent with oxygen saturation< 90% (TS90) on lung cancer mortality and overall mortality | Follow up for 5 years
  A secondary outcome measure in a longitudinal analysis of prospective cohort study.

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea